CLINICAL TRIAL: NCT01873664
Title: Brain Activity During Jaw Tapping Movement in Healthy Subjects and Mild Cognitive Impairment Patients Using Functional Magnetic Resonance Imaging
Brief Title: Functional Magnetic Resonance Imaging Study of Jaw-tapping Movement on Memory Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Seung-Yeon Cho, fellow, Kyung Hee University Hospital at Gangdong, Kyunghee University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NRF-2010-0017278
Record Dates: First submitted 2013-06-03; First posted 2013-06-10 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Memory Disturbances
Keywords: fMRI; Jaw tapping; Memory disorder; Mild cognitive impairment; MCI; Working memory
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Jaw tapping (Experimental): All subjects performed the jaw-tapping for 4 weeks at home.
  Interventions: Behavioral: Jaw-tapping

INTERVENTIONS:
Behavioral: Jaw-tapping — to tap their jaws vertically at 1.6 Hz at home twice a day for 30 seconds every day during four weeks.

SUMMARY:
The purpose of this study is to examine the possibility of using jaw-tapping training as a self-exercise for developing memory and preventing dementia in elderly subjects with memory disturbances using functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
Right-handed female volunteers over the age of 50 years with subjective memory complaints are included in the study. Volunteers with dentures, psychoactive medication, history of stroke, or other neurologic disorders are excluded.

The protocol was approved by the Institutional Review Board of university-based hospital.

After administering the Seoul Neuropsychological Screening Battery (SNSB), Mini-Mental State Examination (MMSE) scores above 24 and Clinical Dementia Rating Scale (CDR) scores of 0 are considered subjective memory complaints (SMC), and MMSE scores above 23 and CDR scores of 0.5 are considered MCI.

All subjects undergo two MRI scans. After the first MRI, the subjects are trained to tap their jaws vertically at 1.6 Hz at home twice a day for 30 seconds every day during four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed female volunteers over the age of 50 years with subjective memory complaints

Exclusion Criteria:

* Volunteers with dentures, psychoactive medication, history of stroke, or other neurologic disorders

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-05; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Brain activity of n-back task | up to 4 weeks
  All subjects perform the jaw-tapping and the n-back memory tasks during blood oxygen level dependent (BOLD) fMRI, before and after practicing the jaw-tapping exercise for 4 weeks at home.
  Pre- and post-test fMRI data during the n-back task are analyzed using statistical parametric maps of brain activation.

SECONDARY OUTCOMES:
Brain activity of jaw-tapping task | baseline and 4 weeks
  All subjects perform the jaw-tapping and the n-back memory tasks during blood oxygen level dependent (BOLD) fMRI, before and after practicing the jaw-tapping exercise for 4 weeks at home.
  Pre- and post-test fMRI data during the jaw-tapping task are analyzed using statistical parametric maps of brain activation.

OTHER OUTCOMES:
Performance scores of the n-back task | baseline and 4 weeks
  One-back task performance of each subject is assessed by analyzing responses obtained during scanning.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Mi Park, Ph.D, Principal Investigator — Professor, Kyung Hee University
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea